CLINICAL TRIAL: NCT00232973
Title: A Prospective, Multi-Centre, Double Blind, Randomized, Placebo Controlled Trial to Evaluate the Safety and Efficacy of ICXP007 in a Phase III Trial With Four-Layer Therapeutic Compression, for the Treatment of Non-Infected Skin Leg Ulcers, Due to Venous-Insufficiency
Brief Title: Safety and Efficacy Study of ICXP007 With Compression Bandaging for the Treatment of Non-Infected Venous Leg Ulcers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intercytex (Industry)
Responsible Party: Intercytex
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-VLU-003
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-02

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ICXP007

SUMMARY:
The main purpose of the study is to compare treatment of non-infected venous leg ulcers using ICXP007 combined with four-layer compression bandaging, placebo combined with four-layer compression bandaging and four-layer compression bandaging alone.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have a graft-ready venous leg ulcer of at least 3 months duration, which has not, responded to standard conventional therapy.
2. Individuals who have an Ankle Brachial Pressure Index (ABPI/ABI) of greater than or equal to 0.8 measured by Doppler sonography.
3. Individuals who have venous incompetency as defined by > 1.0 seconds in vein segments on standing reflux exam by duplex or an abnormal venous refill time of < 21 seconds by PPG or > 2 cc per second by APG. Duplex or PPG/APG will be used to establish venous insufficiency. Doppler will be utilized to rule out arterial disease.
4. Individuals who have a target wound which is between 2 cm2 to 20 cm2 in area at the screening assessment.
5. Individuals who are ambulatory.
6. Individuals who have voluntarily signed and dated a patient IRB/EC approved Informed Consent Form (ICF).
7. Individuals, who are, in the opinion of the Investigator, able to understand this study, co-operate with the study procedures and are willing to return to the clinic for all the required follow-up visits.

Exclusion Criteria:

1. Individuals with a known hypersensitivity to Aprotinin or any other constituents of Tisseel VH S/DTM i.e. Fibrinogen (human), thrombin (human) and Calcium Chloride, Bovine and Porcine products.
2. Individuals who have a haemoglobin or serum albumin level which is < 10 g/dL or < 2.5 g/dL respectively, or is otherwise outside the normal range and deemed clinically significant.
3. Females who are pregnant, lactating, or who have not reached menopause and are not abstinent or practicing an acceptable means of birth control as determined by the Investigator for the duration of the study.
4. Individuals younger than 18 years of age.
5. Individuals with abnormal blood biochemistry defined as 3 times that of the upper limit of the normal range and/or any other abnormal laboratory finding considered clinically significant.
6. Individuals who have exposed bone, tendon or fascia visible around the target wound.
7. Individuals with evidence of collagen vascular diseases, such as vasculitis or rheumatoid arthritis, under active treatment.
8. Individuals with evidence of cellulitis or osteomyelitis during the previous 4 weeks.
9. Individuals who have a target wound which shows signs of clinical infection or who have a wound that has presence of ß-haemolytic streptococcus upon culture, or the Investigator suspects may be severely infected. Individuals may be enrolled upon eradication of the ß-haemolytic streptococcus infection/organism.
10. Individuals who have any clinically significant medical condition that would impair wound healing as determined by the Investigator, including uncontrolled diabetes as determined by HbA1C (>12%), or immune disease.
11. Individuals who are known to abuse alcohol or drugs currently, or to have psychological disorders that could affect follow-up care or treatment outcomes.
12. Individuals who have chronic renal insufficiency requiring haemodialysis.
13. Individuals who have received short course corticosteroids within 30 days, or oral or parenteral chronic immunosupressants within 90 days prior to treatment.
14. Individuals who have, or are suspected of having malignancy, or who have received treatment for any active malignancy, apart from non-melanomatic skin cancer, within 3 months prior to treatment.
15. Individuals who have participated in a clinical study of any investigational product within 2 months prior to treatment.
16. Individuals who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
17. Individuals previously enrolled/randomized in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2005-07

PRIMARY OUTCOMES:
Incidence of 100% closure (epithelialized) at any time during the initial 12 weeks of the treatment period. | 12 weeks

SECONDARY OUTCOMES:
Overall rate of wound area reduction during treatment.
Time to first closure.
Incidence of closure at 16, 20 and 24 weeks.
Incidence of reopening at up to 16, 20 and 24 weeks.
Incidence of re-closure at 16, 20 and 24 weeks.
Qualitative levels of wound pain.
Percentage of Day 0 wound surface area.
Percentage reduction in wound surface area from previous visit.
Percentage reduction in wound surface area from Day 0.
Appearance of new ulcer in the target wound area post closure.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (30):
  - Institute for Advanced Wound Care, Montgomery, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Alameda County Medical Center, Alameda, California
  - Manzainto Medical Clinic, Carmichael, California
  - Bay Area Foot Care, Castro Valley, California
  - M Limova, MD, Fresno, California
  - VA Medical Center, Sacramento, California
  - Bay Area Foot care, San Francisco, California
  - University of Florida, Department of Surgery, Gainesville, Florida
  - Dr Francisco Kerdel, Miami, Florida
  - Doctor's Research Network, Miami, Florida
  - Dermatology and Cosmetic Specialists, Miramar, Florida
  - Dr. Robert Snyder, Tamarac, Florida
  - National Centre for Limb Preservation, Niles, Illinois
  - Centre for Lower Ambulatory Research, Rosalind Franklin University of Medicine & Science, North Chicago, Illinois
  - Prairie Vascular Institute, Springfield, Illinois
  - The Wound Healing Center, Terre Haute, Indiana
  - Boston Medical Center, Department of Vascular Surgery, Boston, Massachusetts
  - Dermatology, PLLC, Ann Arbor, Michigan
  - Advanced Foot and Ankle Center, Las Vegas, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - UNC Wound Care Clinic, Chapel Hill, North Carolina
  - OSU Comprehensive Wound Center, Columbus, Ohio
  - St Vincent Health Center, Erie, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - Penn North Centers for Advanced Wound Care, Warren, Pennsylvania
  - Roger Williams Medical Centre, Providence, Rhode Island
  - Madigan Army Medical Center, Tacoma, Washington
  - Central Washington Podiatry, Yakima, Washington
- Canada (10):
  - Western Canada Dermatology Institute, Edmonton, Alberta
  - Clinical Trials Unit, Skin Care Centre, Vancouver, British Columbia
  - Eastern Canada Cutaneous Research Associates Ltd, Halifax, Nova Scotia
  - Parkwood Hospital, St Joseph's Health Care, London, Ontario
  - Gary Sibbald, MD, Mississauga, Ontario
  - Entralogix, Oakville, Ontario
  - Dermatology Daycare, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Entralogix, Welland, Ontario
  - Centre Medical Ste-Dorothee, Laval, Quebec
- United Kingdom (17):
  - Department of Vascular Surgery, Manchester Royal Infirmary, Manchester, Lancashire
  - Clatterbridge Hospital, Surgical Outpatients, Upton, Wirral
  - Aberdeen Royal Infirmary, Aberdeen
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, University Department of Vascular Surgery, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Cardiff University, Cardiff
  - St Richards Hospital, Chichester
  - Russells Hall Hospital, Dudley
  - Gloucestershire Royal Hospital, Gloucester
  - Hull Royal Infirmary, Hull
  - Vascular Surgical Unit, Leeds General Infirmary, Leeds
  - St George's Hospital, London
  - Derriford Hospital, Plymouth
  - The Willows Centre for Health, Salford
  - Arrowe Park Hospital, Upton
  - Wrexham Maelor Hospital, Wrexham